CLINICAL TRIAL: NCT01047748
Title: A Randomized Clinical Trial of Intra-fetal Versus Intra-amniotic Digoxin Prior to Second-Trimester Pregnancy Termination
Brief Title: A Trial of Digoxin Before Second-Trimester Abortion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: White, Katharine O'Connell, M.D., M.P.H. (Individual)
Collaborators: Society of Family Planning (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 20082058
Record Dates: First submitted 2010-01-11; First posted 2010-01-13 (Estimated); Last update posted 2013-05-01 (Estimated); Status verified 2013-04

CONDITIONS: Induced Abortion
Keywords: abortion
MeSH Terms: interventions — Digoxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- intra-fetal injection (Active Comparator): Subjects will receive an intra-fetal digoxin injection one day prior to their second-trimester surgical abortion
  Interventions: Drug: intra-fetal digoxin injection
- intra-amniotic injection (Active Comparator): Subjects will receive an intra-amniotic digoxin injection one day prior to their second-trimester surgical abortion
  Interventions: Drug: intra-amniotic digoxin injection

INTERVENTIONS:
Drug: intra-fetal digoxin injection — Single transabdominal injection of digoxin 1 mg into the fetus
  Other Names: Lanoxin
  Arms: intra-fetal injection
Drug: intra-amniotic digoxin injection — Single transabdominal injection of digoxin 1 mg into the amniotic fluid
  Other Names: Lanoxin
  Arms: intra-amniotic injection

SUMMARY:
The purpose of our study is to determine the optimum route for the injection of digoxin prior to second-trimester surgical abortion.

DETAILED DESCRIPTION:
Of the 1.2 million abortions each year in the U.S., approximately 12% take place in the second trimester of pregnancy. The preferred technique for second-trimester pregnancy termination is dilation and evacuation, or D&E. In 2006, 144,000 D&Es were performed in the U.S. Clinicians often achieve preoperative fetal asystole by a maternal transabdominal injection of digoxin. Prior to D&E, providers use digoxin to induce fetal death 1) for providers' preference to facilitate surgical delivery of the fetus, and/or 2) for patients who express a desire for fetal death prior to the abortion.

The use of digoxin to achieve preoperative fetal asystole is widespread, yet there are no evidence-based standards for how to best achieve fetal asystole prior to D&E. Digoxin has been administered by intracardiac, intrathoracic, intrafetal and intra-amniotic routes, with doses varying from 0.25 to 2mg. Clinicians who use digoxin usually inject it one to two days before the D&E. Only one study has assessed the effectiveness of digoxin at varying dosages ; this was a retrospective and nonrandomized analysis. Published failure rates are based on small numbers of patients and are therefore imprecise. Intrafetal digoxin injection may be more effective, but is a technically more difficult procedure than intra-amniotic injection. The pharmacodynamics of digoxin when used for feticide are also unknown. The objective of this study is to determine the optimum route for digoxin injection (intrafetal or intra-amniotic) that will maximize patient safety while maintaining effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years old
* English or Spanish speaking
* be able to give informed consent
* documented fetal cardiac activity.

Exclusion Criteria:

* significant medical illness or cardiovascular disease
* current use of cardiac or antihypertensive medications
* cardiac arrhythmia on preoperative EKG
* multiple gestation
* morbid obesity (BMI greater than 40)
* known digoxin allergy

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 272 (Actual)
Dates: Start 2011-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
difference in fetal asystole rates between groups | one day

SECONDARY OUTCOMES:
digoxin-related side effects | one day
differences in surgical procedure between groups | one day
subject satisfaction | one day
serum digoxin levels in study subgroup | one day

CONTACTS AND LOCATIONS:
Overall Officials: Katharine O White, MD, MPH, Principal Investigator — Physicians for Reproductive Choice and Health
Locations (1):
- Planned Parenthood Los Angeles - Bixby Health Center, Los Angeles, California, United States

REFERENCES:
- [Background] Jackson RA, Teplin VL, Drey EA, Thomas LJ, Darney PD. Digoxin to facilitate late second-trimester abortion: a randomized, masked, placebo-controlled trial. Obstet Gynecol. 2001 Mar;97(3):471-6. doi: 10.1016/s0029-7844(00)01148-0. PMID 11239659
- [Background] Molaei M, Jones HE, Weiselberg T, McManama M, Bassell J, Westhoff CL. Effectiveness and safety of digoxin to induce fetal demise prior to second-trimester abortion. Contraception. 2008 Mar;77(3):223-5. doi: 10.1016/j.contraception.2007.10.011. Epub 2008 Jan 22. PMID 18279695
- [Background] Drey EA, Thomas LJ, Benowitz NL, Goldschlager N, Darney PD. Safety of intra-amniotic digoxin administration before late second-trimester abortion by dilation and evacuation. Am J Obstet Gynecol. 2000 May;182(5):1063-6. doi: 10.1067/mob.2000.105438. PMID 10819828
- [Derived] White KO, Nucatola DL, Westhoff C. Intra-fetal Compared With Intra-amniotic Digoxin Before Dilation and Evacuation: A Randomized Controlled Trial. Obstet Gynecol. 2016 Nov;128(5):1071-1076. doi: 10.1097/AOG.0000000000001671. PMID 27741192